CLINICAL TRIAL: NCT01763385
Title: Erlotinib With Concurrent Brain Radiotherapy and Secondary Brain Radiotherapy After Recurrence With Erlotinib in NSCLC Non-increased-intracranial-pressure Symptomatic Brain Metastases: A Prospective Multicenter Trial(TRACTS)
Brief Title: Erlotinib With Concurrent Brain Radiotherapy and Secondary Brain Radiotherapy After Recurrence With Erlotinib in NSCLC Non-increased-intracranial-pressure Symptomatic Brain Metastases
Acronym: TRACTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wu Jieping Medical Foundation (Other)
Collaborators: Fudan University (Other); Changhai Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Longhua Hospital (Other); RenJi Hospital (Other); Shanghai Armed Police Hospital (Unknown); Shanghai Chest Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yang Huan Jun, Fudan University, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-75-634
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Non-small-cell Lung Cancer; Brain Metastases
Keywords: Erlotinib; brain radiotherapy; NSCLC; brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib & secondary brain radiotherapy (Experimental): Erlotinib until brain tumor progression, then given brain radiotherapy, and continued to take Erlotinib till extracranial lesions progression.
  Interventions: Drug: Erlotinib; Radiation: secondary brain radiotherapy
- Erlotinib & concurrent brain radiotherapy (Other): Erlotinib with concurrent brain radiotherapy, and continued to take Erlotinib after radiotherapy until recurrence or termination for other reasons
  Interventions: Drug: Erlotinib; Radiation: concurrent brain radiotherapy

INTERVENTIONS:
Drug: Erlotinib
Radiation: concurrent brain radiotherapy
  Arms: Erlotinib & concurrent brain radiotherapy
Radiation: secondary brain radiotherapy
  Arms: Erlotinib & secondary brain radiotherapy

SUMMARY:
This project is aim to explore non-increased-intracranial-pressure symptomatic brain metastases of NSCLC, and if the OS of secondary brain radiotherapy after recurrence with Erlotinib is better than Erlotinib with concurrent brain radiotherapy. Treatment group are treated with Erlotinib until brain tumor progression, then gave brain radiotherapy, and continued to take Erlotinib till extracranial lesions progression. Control group are Erlotinib with concurrent brain radiotherapy, and continued to take Erlotinib after radiotherapy until recurrence or termination for other reasons.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years old;
2. Tissue or cell pathological diagnosis of NSCLC;
3. Brain CT or MR validated BM;
4. Non-increased-intracranial-pressure symptomatic BM;
5. Haven't received TKI target treatment;
6. Haven't received brain radiotherapy;
7. Patients in initial treatment should be detected EGFR mutation;
8. Expected survival more than 6 months;
9. KPS no less than 70, or KPS less than 70 caused by paralysis due to recent brain metastases;
10. Liver and kidney function requirements: SGOT/SGPT≦2.5 times of the upper limit, Total bilirubin≦1.5 times of the upper limit, serum Creatinine≦1.5 times of the upper limit;
11. Routine blood test requirements: WBC≧3.0×109/L, NE≧1.8×109/L, PLT≧90×109/L，no requirement for Hb;
12. Blood glucose requirements: within the normal range, diabetic patients are receiving treatment and their glucose was being controlled in a steady state;
13. Female patients in childbearing age: HCG (-);
14. Patients signed an inform Consent.

Exclusion Criteria:

1. Those with Erlotinib drug allergies;
2. Those with mathematical understanding of the most simple life questions, such as "walking", those difficult for doctors to communicate;
3. Those without guardians or families;
4. Those with abnormal routine blood test, liver and kidney function, and blood glucose beyond the above boundaries and difficult to correcting for more than 2 weeks;
5. Those with any unstable medical status (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction (within one year before treatment initiation), and severe arrhythmia, liver, kidney or metabolic disease requiring drug therapy);
6. Those with any other disease, neurological or metabolic dysfunction, and physical examination or laboratory test results showed that the study drugs may increase the risk of treatment-related complications;
7. Pregnant women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3.5year

CONTACTS AND LOCATIONS:
Overall Officials: Huanjun Yang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China